CLINICAL TRIAL: NCT01670604
Title: The Use of Two Modern Hydroxyethyl Starch Solutions in Major Urological Procedures: Effect on Acid-Base Status and Renal Functions
Brief Title: Use of Two Modern Hydroxyethyl Starch Solutions in Major Urological Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mukhtar, Assistant professor of anesthesia Cairo University, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: KAH012
Record Dates: First submitted 2012-08-05; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Urologic Surgical Procedures
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VOL group (Experimental): patients will receive 6% HES 130/0.4 in NaCl 0.9% (Voluven, Fresenius Kabi, Bad Hom-bourg, Germany)
  Interventions: Drug: 6% HES 130/0.4 in NaCl 0.9% (Voluven, Fresenius Kabi, Bad Hom-bourg, Germany)
- TET group (Experimental): patient will receive 6% HES 130/0.42 in a balanced electrolyte containing Na+140 mmol/L, Cl- 118 mmol/L, K +4 mmol/L, Ca++ 2.5 mmol/L, Mg++ 1 mmol/L, acetate- 24 mmol/L and malate-- 5 mmol/L
  Interventions: Drug: Tetraspan, B. Braun, Melsungen, Germany

INTERVENTIONS:
Drug: 6% HES 130/0.4 in NaCl 0.9% (Voluven, Fresenius Kabi, Bad Hom-bourg, Germany)
  Arms: VOL group
Drug: Tetraspan, B. Braun, Melsungen, Germany
  Arms: TET group

SUMMARY:
This study compares the effect of infusion of two types of modern hydroxyethyl starch on the renal function and acid-base in patients undergoing urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age group above 18 years,
* ASA І and ІІ,
* Patients who will be scheduled to undergo radical prostatectomy or cystectomy with bladder replacement

Exclusion Criteria:

* A known allergy to HES,
* Renal insufﬁciency (serum creatinine of >2.5 mg/dL),
* Signiﬁcant hepatic disease (liver function tests more than three times the upper limit of normal),
* Coagulation disorders (INR > 1.5).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Intraoperative volume replacement therapy | From randomization, for the duration of surgery and up to transfer from the operating room to the ICU or recovery room, an expected average of 6 hours
  volume of the study drug in milliliters that will be needed for hemodynamic stabilization until the end of surgery (ie, the cumulative volume of the study drug in milliliters administered up to this time point).

SECONDARY OUTCOMES:
Acid base and Renal function | 24 hours after randomization
  differences in the plasma creatinine concentrations and acid-base homeostasis among the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Hospital, Cairo, Egypt

REFERENCES:
- [Background] Kluft C, Jenks RL, Astrup T. Production of plasminogen actovatpr activity in factor XII-deficient plasma. Thromb Res. 1977 May;10(5):759-64. doi: 10.1016/0049-3848(77)90058-5. No abstract available. PMID 18813
- [Background] Takayanagi I, Maruyama M, Takagi K. Beta-adrenoceptors in the guinea pig treated with egg-albumin. Jpn J Pharmacol. 1977 Apr;27(2):314-6. doi: 10.1254/jjp.27.314. No abstract available. PMID 18633
- [Background] Mitchell AR, Erickson BW, Ryabtsev MN, Hodges RS, Merrifield RB. Tert-butoxycarbonylaminoacyl-4-(oxymethyl)-phenylacetamidomethyl-resin, a more acid-resistant support for solid-phase peptide synthesis. J Am Chem Soc. 1976 Nov 10;98(23):7357-62. doi: 10.1021/ja00439a041. No abstract available. PMID 10319
- [Background] Birke ER. [On the action of antihypotensive agents in sympathicotonic orthostatic hypotension in geriartric patients: comparison between placebo and etilefrin (author's transl)]. Med Klin. 1977 Oct 14;72(41):1696-702. German. PMID 21345